CLINICAL TRIAL: NCT05579366
Title: Phase 1/2 Study of Rina-S in Patients With Locally Advanced and/or Metastatic Solid Tumors
Brief Title: Rinatabart Sesutecan (Rina-S, PRO1184, GEN1184) for Advanced Solid Tumors (GCT1184-01/ PRO1184-001)
Acronym: RAINFOL-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1184-01; CTR20230813 (Registry Identifier: Chinadrugtrials.org.cn); PRO1184-001 (Other: Other Sponsor Identifier); jRCT2051250094 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-10-04; First posted 2022-10-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: High Grade Epithelial Ovarian Cancer; High Grade Serous Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer; Endometrial Cancer; Non-small Cell Lung Cancer; Epidermal Growth Factor Receptor (EGFR)-Mutated Non-Small Cell Lung Cancer (NSCLC); Mesothelioma; Breast Adenocarcinoma; Triple Negative Breast Cancer; Hormone Receptor-positive/Her2 Negative Breast Cancer; Platinum-resistant Ovarian Cancer (PROC); Platinum Sensitive Ovarian Cancer (PSOC); Primary Refractory Ovarian Cancer; Uterine Cancer
Keywords: antibody-drug conjugate; folate receptor alpha; folate receptor; solid tumor; ovarian cancer; primary peritoneal carcinoma; fallopian tube cancer; endometrial cancer; non-small cell lung cancer; mesothelioma; breast cancer; triple negative breast cancer; hormone receptor-positive (HR+)/human epidermal growth factor receptor 2 negative (HER2-) breast cancer; topoisomerase I inhibitor; PROC; epidermal growth factor receptor (EGFR)-mutated NSCLC
MeSH Terms: conditions — Fallopian Tube Neoplasms; Endometrial Neoplasms; Carcinoma, Non-Small-Cell Lung; Mesothelioma; Triple Negative Breast Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Breast Neoplasms | interventions — Carboplatin; Bevacizumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A, B, C, F, G, H, I, J and K (Experimental): Rina-S monotherapy in Part A and at the recommended dose in Parts B, C, F, G, H, I, J and K.
  Interventions: Drug: Rina-S
- Part D1 (Experimental): Rina-S in combination with carboplatin
  Interventions: Drug: Rina-S; Drug: Carboplatin
- Part D2 and I (Experimental): Rina-S in combination with bevacizumab
  Interventions: Drug: Rina-S; Drug: Bevacizumab
- Part D3 and D4 (Experimental): Rina-S in combination with pembrolizumab
  Interventions: Drug: Rina-S; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Rina-S — Intravenous infusion of Rina-S
  Other Names: PRO1184; Rinatabart sesutecan; GEN1184
Drug: Carboplatin — Carboplatin intravenous infusion
  Arms: Part D1
Drug: Bevacizumab — Bevacizumab intravenous infusion
  Arms: Part D2 and I
Drug: Pembrolizumab — Pembrolizumab intravenous infusion
  Arms: Part D3 and D4

SUMMARY:
This study will test the safety, including side effects, and determine the characteristics of a drug called Rina-S in participants with solid tumors.

Participants will have solid tumor cancer that has spread through the body (metastatic) or cannot be removed with surgery (unresectable).

DETAILED DESCRIPTION:
This is a Phase 1/2 study of Rina-S; also known as GEN1184, formerly known as PRO1184, a folate receptor alpha (FRα) targeted antibody-drug conjugate, to evaluate the safety, tolerability, pharmacokinetics (PK), and antitumor activity of Rina-S in participants with selected locally advanced and/or metastatic solid tumors, including epithelial ovarian cancer, endometrial cancer, breast cancer, non-small cell lung cancer, and mesothelioma.

The study consists of multiple parts:

Part A: monotherapy cohorts

Part B: tumor-specific monotherapy dose-expansion cohorts

Part C: platinum-resistant ovarian cancer (PROC) monotherapy cohort

Part D: combination therapy cohorts

Parts F and G: a monotherapy endometrial cancer (EC) cohort

Part H: a monotherapy PROC cohort

Part I: platinum-sensitive ovarian cancer (PSOC) cohort

Part J: a monotherapy PROC cohort

Part K: a monotherapy high-grade ovarian cancer cohort

Participants will continue to receive study treatment until the first instance of disease progression, unacceptable toxicity, investigator decision, consent withdrawal, study termination by the Sponsor, pregnancy, or death.

ELIGIBILITY:
Inclusion Criteria:

Part A and B:

* Histologically or cytologically confirmed metastatic or unresectable solid malignancy including ovarian cancer (must have epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer), endometrial cancer, non-small cell lung cancer (Part A), EGFR-mutated NSCLC (Part B), breast cancer (hormone receptor positive, HER2-negative and triple-negative) (Part A), mesothelioma or cervical cancer (Part B).
* Previously received therapies known to confer clinical benefit.
* Measurable disease per RECIST v1.1 for all tumor types other than pleural mesothelioma which will use mRECIST v1.1 at baseline.

Part C and H:

Participants must have histologically or cytologically confirmed metastatic or unresectable epithelial ovarian cancer as specified below.

* High grade serous ovarian cancer, primary peritoneal cancer, or fallopian tube cancer (excluding endometrioid, clear cell carcinomas, mucinous, low grade, and those with a sarcomatous or neuroendocrine element)
* Participants must have received up to 3 prior lines of therapy. Participants may have had up to to 4 prior lines of therapy are allowed if MIRV is locally approved and was used as the last line of therapy. Participants must have progressed radiographically on or after their most recent line of therapy.
* Participants must have platinum-resistant ovarian cancer.
* Participants must have received prior bevacizumab or approved biosimilar.
* Participants with known or suspected deleterious germline or somatic BRCA mutations (as determined by Food and Drug Administration [FDA]-approved test in a Clinical Laboratory Improvement Amendments [CLIA]-certified laboratory; or locally approved equivalent) and who achieved a complete or partial response to platinum-based chemotherapy must have been treated with a poly ADP-ribose polymerase (PARP) inhibitor as maintenance treatment.
* Measurable disease per the RECIST v1.1 at baseline.

Part D:

Cohort D1:

* Participants must have platinum-sensitive ovarian cancer.
* Participants must have received 1 to 3 prior lines of therapy.

Cohort D2:

* Participants must have primary platinum-refractory, platinum-resistant, or platinum-sensitive ovarian cancer.
* Participants with primary platinum-refractory ovarian cancer must have received ≤2 prior lines of therapy. Primary platinum-refractory ovarian cancer is defined as a lack of response or by progression within 91 days after completing front-line platinum containing therapy.
* Participants must have received 1 to 3 prior lines of therapy for platinum-resistant ovarian cancer (PROC), and up to 4 prior lines of therapy for platinum-sensitive ovarian cancer (PSOC). Prior treatments may have included bevacizumab, PARP inhibitor, and MIRV.

  * Participants with PSOC must have disease progression on or after maintenance treatment, or at least 6 months (>183 days) or more from the last dose of platinum-based therapy.

Cohort D3 and D4:

• Endometrial cancer (any subtype excluding sarcoma).

Part F and G:

* Participants must have histologically or cytologically confirmed EC.
* Recurrent progressive EC (any subtype excluding neuroendocrine tumors, carcinosarcoma, or endometrial sarcoma) following prior therapy.
* Participants must have received 1 to 3 prior lines of therapy, and must have progressed radiographically on or after their most recent line of therapy:
* Participants must have received prior platinum-based chemotherapy and a programmed death-ligand 1 (PD-[L])1 inhibitor.
* Participants who progress >12 months after completion of prior adjuvant or neoadjuvant platinum-based chemotherapy must receive 1 additional cytotoxic systemic treatment prior to enrollment in this study.
* Hormonal therapy alone (i.e., without chemotherapy) will not be counted as a separate line of therapy.
* Measurable disease per the RECIST Version 1.1 at baseline.

Part I:

* Participants must have histologically or cytologically confirmed high grade serous or endometrioid epithelial ovarian cancer, fallopian tube cancer and primary peritoneal cancer (excluding clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of the above histologies or low grade/borderline ovarian tumors).
* Participants must have platinum sensitive ovarian cancer.
* Measurable disease per the RECIST Version 1.1 at baseline.

Part J:

* Participants must have high grade epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer including serous, endometrioid, and clear cell carcinomas, and excluding mucinous, low grade, and those with a sarcomatous or neuroendocrine element.
* Measurable disease per the RECIST Version 1.1 at baseline.

Part K:

* Participants must have histologically or cytologically confirmed metastatic or unresectable ovarian cancer (must have high grade epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer including serous, endometrioid, and clear cell carcinomas, and excluding mucinous, low grade, and those with a sarcomatous or neuroendocrine element).
* Participants must have primary platinum-refractory, platinum-resistant, or platinum-sensitive ovarian cancer.
* Measurable disease per the RECIST Version 1.1 at baseline.

Exclusion Criteria:

* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids within the past 2 years, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Prior therapy with a topoisomerase 1 inhibitor-based antibody drug conjugate.

Note: Other protocol-defined inclusion/exclusion may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 764 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Parts A, B, and D - Incidence of Treatment-Emergent Adverse Events (TEAEs) [Safety and Tolerability] | Through end of treatment, up to approximately 1 year.
Parts A, and D - Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (each cycle is 21 days)
  The proportion of participants experiencing DLT.
Parts C, F, G, H, I, and J- Objective Response Rate (ORR) as Assessed by Blinded Independent Central Review (BICR, Parts C, E, and F) or Investigator (Part G, I, and J) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Through end of treatment, up to approximately 1 year.
  Participants who achieve partial response (PR) or complete response (CR) per RECIST v1.1 criteria.
Part K (US Participants Only) - Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Findings by Holter | Cycles 1 to 3 (each cycle is 21 days)

SECONDARY OUTCOMES:
Parts A, B, and D - Best Overall Response (BOR) | Up to approximately 1 year.
  Participants who achieve CR or PR. Best response as assessed by the investigator per RECIST v1.1 criteria for all tumor types other than pleural mesothelioma which will use modified RECIST (mRECIST) v1.1.
Parts A, B, and D - ORR | Up to approximately 1 year.
  Participants who achieve PR or CR per RECIST v1.1 criteria.
Parts A, B, and D - Disease Control Rate (DCR) | Up to approximately 1 year.
  Participants who achieve stable disease, PR or CR per RECIST v1.1 criteria.
Parts A, B, C, D, F, G, H, I, and J - Progression-Free Survival (PFS) | Through end of treatment, up to approximately 1 year.
  Time from start of treatment to first documented disease progression or death
Parts C, F, G, H, I and J - Overall survival (OS) | Up to approximately 2 years.
  Time from the start of study treatment to the date of death from any cause
Parts A, B, C, D, F, H, I and J - Duration of Objective Response (DOR) | From date of enrollment until the date of first documented disease progression or date of study withdrawal, whichever came first, assessed up to 12 months.
  Time from the first documentation of an objective tumor response (CR or PR) to the first documented tumor progression or death
Parts A, B, and D - Peak Plasma Concentration (Cmax) for Rina-S | Through end of treatment, up to approximately 1 year.
  Measurement of maximum plasma concentration after the administration of Rina-S.
Parts A, B, and D - Area Under the Plasma Concentration Versus Time Curve (AUC) for Rina-S | Through end of treatment, up to approximately 1 year.
  Measurement of AUC after the administration of Rina-S.
Parts A, B, and D -Time to Reach Cmax (Tmax) for Rina-S | Through end of treatment, up to approximately 1 year
Parts A, B, and D - Trough Concentrations (Ctrough) for Rina-S | Through end of treatment, up to approximately 1 year
Parts A, B, and D - Apparent Terminal Half-life (t1/2) for Rina-S | Through end of treatment, up to approximately 1 year
Parts C, D, H and J - CA-125 Response Determined Using the Gynecologic Cancer Intergroup (GCIG) Criteria | Through end of treatment, up to approximately 1 year
Parts C, F, H, I, J, and K - Number of Participants with Type, Incidence, Severity, Seriousness as per Common Terminology Criteria for Adverse Events (CTCAE) v5.0, and Relatedness of Adverse Events (AEs) | Through end of treatment, up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (67):
- United States (37):
  - USOR HonorHealth, Phoenix, Arizona
  - USOR Arizona Oncology Associates, Tucson, Arizona
  - University of California Los Angeles Medical Center, Los Angeles, California
  - University of California, San Diego; Moores Cancer Center, San Diego, California
  - USOR Sansum Clinic, Santa Barbara, California
  - Providence Medical Foundation, Santa Rosa, California
  - USOR Florida Cancer Specialists South, Fort Myers, Florida
  - USOR Florida Cancer Specialists North, St. Petersburg, Florida
  - USOR Florida Cancer Specialists East, West Palm Beach, Florida
  - Augusta University Georgia Cancer Center, Augusta, Georgia
  - University of Kansas Medical Center (KUMC), Westwood, Kansas
  - USOR Maryland Oncology Hematology, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - USOR Minnesota Oncology Hematology, Maplewood, Minnesota
  - MD Anderson Cancer Center at Cooper- Two Cooper Plaza, Camden, New Jersey
  - Ohio State University Comprehensive Cancer Center (OSUCCC)- The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - University of Oklahoma - Health Sciences Center, Oklahoma City, Oklahoma
  - USOR Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Compass Oncology - Rose Quarter, Portland, Oregon
  - USOR Alliance Cancer Specialist, Doylestown, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - USOR Texas Oncology, Abilene, Texas
  - Texas Oncology - Central / South Texas, Austin, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - USOR Texas Oncology, Fort Worth, Texas
  - Texas Oncology - Northeast TX, Tyler, Texas
  - USOR Texas Oncology Gulf Coast, Woodland, Texas
  - START Mountain Region, West Valley City, Utah
  - USOR Virginia Cancer Specialists, Fairfax, Virginia
  - USOR Virginia Oncology Associates, Norfolk, Virginia
  - Swedish Cancer Institute, Seattle, Washington
- China (20):
  - Cancer hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Hunan Cancer Hospital - Phase 1, Changsha, Hunan
  - Hunan Cancer Hospital - Thoracic Medicine Dept II, Changsha, Hunan
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Obstetrics & Gynecology Hospital of Fudan University, Chengdu, Shanghai Municipality
  - Fudan University Shanghai Cancer Center - Gynecologic Oncology, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center- Phase 1, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Shanghai, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Fujian Cancer Hospital, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangdong
  - Second Affiliated Hospital of Zhengzhou University, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Hubei
  - Second Hospital of Shanxi Medical University, Shanxi
  - Shanxi Cancer Hospital, Shanxi
  - Liaoning Cancer Hospital & Institute, Shengyang
  - Tianjin Cancer Hospital, Tianjin
- Japan (10):
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Saitama Medical University-International Medical Center, Hidaka, Saitama
  - Shizuoka Cancer Center, Nagaizumi-chō, Shizuoka
  - Cancer Institute Hospital of JFCR, Koto, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No